CLINICAL TRIAL: NCT04811742
Title: Effect of Immersion Bathing and Showering Applications on Comfort Level and Physiological Parameters of Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Gülzade Uysal, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 010
Record Dates: First submitted 2021-03-12; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Preterm Birth
Keywords: Immersion bathing; showering; comfort; physiological parameters
MeSH Terms: conditions — Premature Birth | interventions — Baths

STUDY DESIGN:
Intervention Model Description: A power analysis was performed to determine the sample size, which was calculated to include 31 newborns for each study group under the conditions of 0.05 significance level, 0.95 confidence interval and 0.95 power. Due to possible missing data, the sample size was increased by 10%, and the study was completed with a total of 69 newborns, including 35 in the immersion bathing group and 34 in the showering group.In this study, randomization by throwing a dice was used to allocate newborns into study groups. A dice was rolled for each newborn who met the study inclusion criteria, whereby the newborn was assigned to the immersion bathing group when an even number was observed, and to the showering group when an odd number was observed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immersion bathing group (Experimental): Immersion bathing was started by placing the baby's whole body, except for the head and neck, into a bathtub of warm water with a depth of 13-14 cm. The baby was shampooed and cleaned in the tub. Then, the baby was taken out of the water and rinsed over the tub. Finally, the baby was wrapped with a towel, taken to the radiant and dried, thus the process of bathing was completed.
  Interventions: Other: bathing
- showering group (Experimental): Shower was started by keeping the baby's face down and firmly gripping the baby from his/her armpit and head by one of the nurse's hands. The baby was washed under running water with the other hand. The second nurse assisted to ensure the flow of water. After the baby was rinsed, he/she was wrapped with a towel, taken to the radiant and dried, thus the process of bathing was completed.
  Interventions: Other: bathing

INTERVENTIONS:
Other: bathing — immerson bathing and showering

SUMMARY:
Effect of immersion bathing and showering applications on comfort level and physiological parameters of Newborn

DETAILED DESCRIPTION:
This study aims to determine the effect of immersion bathing and showering on comfort levels and physiological parameters of newborns in neonatal intensive care units.

This is a randomized controlled experimental study. The sample consisted of a total of 69 newborns who were born at the 37th gestational week and above, were referred to the neonatal intensive care unit of a training and research hospital, and met the study inclusion criteria. Study groups were determined through randomization by throwing a dice (immersion bathing group:35, showering group:34). Environmental variables were kept the same for both groups. Physiological parameters (respiration, high heart rate, oxygen saturation, body temperature) and comfort levels of newborns in both groups were compared before, just after and 15 minutes after the bath. Their comfort levels were measured using the Newborn Comfort Behavior Scale (NCBS).

ELIGIBILITY:
Inclusion Criteria:

* Being a newborn born at the 37th gestational week and above,
* Completing 24 hours following the birth
* Having a stable condition (no tachycardia and bradycardia)

Exclusion Criteria:

* Having respiratory failure and distress (having respiratory rate between 30-60, not being monitored in the ventilator, having oxygen saturation of 90% and above, having no need for high concentrations of oxygen via methods such as Hood and CPAP)
* Having signs of infection, fever and hypothermia (having an ideal body temperature between 36-37.3 ℃)
* Having neurological problems (hypotonia, hypertonics, etc.), no history of convulsions, using no sedative medication, and having a normal cranial USG.

Ages: 37 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — newborn
Enrollment: 69 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Newborn Comfort Behavior Scale (NCBS) | 2 minute
  The scale was developed by Dijk et al. (2009), and its Turkish validity and reliability study was performed by Kahraman et al. (2014). This is a five-point Likert type scale with six factors: alertness, calmness/agitation, respiratory response, physical movement, crying, muscle tone, and facial tension. The NCBS is used by nurses to assess the baby's comfort, pain and distress. Total score ranges from 6 to 30. A lower score indicates a higher newborn comfort level. A total score between 9-13 indicates that the baby is "comfortable", whereas a total score between 14-30 indicates that the baby has pain and distress, that is, is "uncomfortable" and needs comfort enhancing interventions.
Respiratory rate | 1 minute
heart rate | 1 minute
oxygen saturation | 1 minute
body tempreture | 1 minute

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No